CLINICAL TRIAL: NCT06803381
Title: Somesthesia in Cancer Patients: Variability and Influence on Eating Experience
Acronym: SOMEST'ALIM2
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0539; 2024-A02687-40 (Other: ID-RCB)
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Digestive Cancers; Breast Cancer; Gynecologic Cancer; Lung Cancer; Nose Cancer; Throat Cancer; Ear Cancer
Keywords: Cancer; nutrition; somesthesia; food; perceptions
MeSH Terms: conditions — Gastrointestinal Neoplasms; Breast Neoplasms; Lung Neoplasms; Nose Neoplasms; Ear Neoplasms; Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Before food testing patients will perform a saliva test in order to determine their saliva quality and quantity. A Saliva-Check BUFFER kit will be used and visual hydration, saliva consistency, pH, volume and buffering capacity will be examined. Results will be available immediately, so it won't be necessary to proceed to a biological storage or laboratory analyses. Thus, samples will be discarded immediately after the test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with cancer and under treatment from at least two months.: The study will involve adult subjects with different types of cancer (digestive, gynecological, breast, ENT, lung) receiving active anticancer treatment (chemotherapy, targeted therapy, immunotherapy, etc., except patients undergoing ENT radiotherapy) in a standard of care program. Patients participating to the trial will perform a salivary test, an evaluation of the sensory capacity, food tasting and will answer to different questionnaires
  Interventions: Other: Salivary test; Other: Food tasting; Other: Questionnaires; Other: sensory capacity evaluation

INTERVENTIONS:
Other: Salivary test — In order to determine the quantity and quality of patients saliva before food tasting a saliva test will be performed using a Saliva-Check BUFFER kit. A small quantity of saliva will be collected and discarded immediately after the test result obtained.
  The test will be done only once for each patient.
Other: Food tasting — Patients will be invited to taste four different food samples, 2 sweet and 2 salty samples, and to evaluate them using a visual analog scale (0 : I don't like at all to 100 : I like a lot). The intervention will be done once for each patient during one of their standard of care treatment visit.
Other: Questionnaires — Patients will be invited to answer to some questionnaires : socio-demographics, appreciation of food samples, self-assessment of oral symptoms and sensory perceptions, QLQ-C30 quality of life and food quality of life questionnaire. They will answer to all questionnaires only once during participation to the study.
Other: sensory capacity evaluation — For the sensory capacity the test 6-n-propylthiouracil (PROP) taste strip will be used. One tasting strip will be placed on the tongue and patients will be asked to assess the intensity of bitterness.
  The test will be done only once for each patient.

SUMMARY:
Patients with cancer are at high risk of denutrition, in France 39% of these patients suffer of malnutrition. This can affect the immunity, the mental balance and impact the treatment response and the quality of life.

Cancer treatments cause many side effects related to food intake as well as sensory alteration, important factor contributing to reduced appetite and inadequate food intake to cancer patients.

SOMEST'ALIM2 is a prospective, non-randomized, monocentric, multisite study that aims to evaluate the appreciation of patients with different types of cancer (digestive, gynecological, breast, ear, nose and throat (ENT) or lung) of two different food versions (sweet and salty), in standard and enhanced version.

Patients must be under treatment from at least two months, and before food testing their sensory capacity and quantity and the quality of their saliva will be tested. They will also be asked to answer to different questionnaires: socio-demographics, appreciation of food samples, self-assessment of oral symptoms and sensory perceptions, MD, Quality of Life Questionnaire (QLQ-C30) and food quality of life questionnaire.

In a context of sensory alterations patients should appreciate more the enhanced food versions. Patients perception of food will be evaluated using a visual analogue scale and results will be correlated with saliva characteristics, subjective sensory perceptions and oral symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 70 years old
* Patient with digestive, breast, gynecologic, ENT or lung cancer
* Patient receiving a cancer treatment from at least two months
* Patient having given his free, informed and express written consent

Exclusion Criteria:

* Patient having a radiotherapy treatment for an ENT cancer
* Patient with a known food allergy/intolerance to food samples (which may contain dairy products)
* Patient unable to swallow soft food
* Patient having presented nausea and vomiting during the last 24 hours
* Patient with severe inflammation of the mouth or throat (ulcers, mucus)
* Patient with cognitive disorders and memory loss
* Pregnant women or breastfeeding
* Adult under legal protection (guardianship)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with different types of cancer: digestive, breast, gynecologic, ENT, lung and aged between 18 and 70 years.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2025-03-13 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale (VAS) score | Day 1
  The score difference of a visual analogue scale (VAS) (0 : I don't like at all to 100 : I like a lot) will be used to evaluate perception of patients with cancer on two different versions of food. The scale unit will be in mm and the difference in VAS score between the two food categories will be compared (hedonic delta).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Amandine BRUYAS, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Service d'Oncologie Médicale - Hôpital de jour Hôpital Edouard Herriot, Lyon
  - Service d'Oncologie Médicale - Hôpital de jour Hôpital de la Croix Rousse, Lyon

IPD SHARING:
Plan to Share IPD: Undecided